CLINICAL TRIAL: NCT06937047
Title: Efficacy and Safety of Cold Versus Hot Snare Polypectomy for Removal of 4-10 mm Pedunculated Colorectal Polyps: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Cold Versus Hot Snare Polypectomy for Removal of 4-10 mm Pedunculated Colorectal Polyps
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Clinical Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202504
Record Dates: First submitted 2025-04-17; First posted 2025-04-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold snare polypectomy group (Experimental)
  Interventions: Procedure: cold snare polypectomy
- hot snare polypectomy group (Active Comparator)
  Interventions: Procedure: hot snare polypectomy

INTERVENTIONS:
Procedure: cold snare polypectomy — Cold snare polypectomy was conducted for the removal of 4-10 mm pedunculated colorectal polyps.
  Arms: cold snare polypectomy group
Procedure: hot snare polypectomy — Hot snare polypectomy was conducted for the removal of 4-10 mm pedunculated colorectal polyps.
  Arms: hot snare polypectomy group

SUMMARY:
This was a non-inferiority randomized controlled trial designed to compare the efficacy and safety of cold versus hot snare polypectomy for the removal of 4-10 mm pedunculated colorectal polyps. The primary outcome was delayed postpolypectomy bleeding. The secondary outcomes included immediate postpolypectomy bleeding, procedure time, en bloc resection, complete histologic resection, use of haemostatic clips and perforation rate.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old, male and female
2. Proposed colonoscopy and colonoscopy detection of at least one 4-10 mm pedunculated colorectal polyp

Exclusion Criteria:

1. Contraindication to colonoscopy or polypectomy
2. Use of antiplatelet or anticoagulant drugs within 1 week before polypectomy
3. Alarming signs and symptoms of colorectal cancer (blood in stool, black stool, unexplained anaemia and weight loss, abdominal mass, positive rectal examination; or imaging and laboratory tests highly suspicious for colorectal cancer) or endoscopic manifestations of polyps highly suspicious for high-grade intraepithelial neoplasia or carcinoma
4. Comorbidity with inflammatory bowel disease, colonic polyposis, or active gastrointestinal bleeding
5. Inadequate bowel preparation
6. Pregnant or lactating women
7. Failure to sign the informed consent form
8. Patients deemed ineligible by investigators to enrol in the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
delayed postoperative bleeding | interviewed by telephone on days 2 and 14 after polypectomy
  bleeding that developed within 2 weeks after the patient left the endoscopy unit

SECONDARY OUTCOMES:
immediate postpolypectomy bleeding | during the polypectomy
  Blood spray or persistent oozing for more than 60 seconds requiring endoscopic intervention
procedure time | during the polypectomy
  The duration from the appearance of the snare on the monitor to the time when the endoscope was withdrawn from the lesion
en bloc resection | during the polypectomy
  Removal of a polyp with a single cut and was assessed by the colonoscopist
complete histologic resection | during the polypectomy
  Clear resection margins, no polyp involvement
use of haemostatic clips | during the polypectomy
perforation rate | during the polypectomy, and interviewed by telephone on days 2 and 14 after polypectomy
  Proportion of patients with intraoperative or postoperative perforation

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arimoto J, Chiba H, Tachikawa J, Yamaoka K, Yamazaki D, Higa A, Okada N, Suto T, Kawano N, Niikura T, Kuwabara H, Nakaoka M, Ida T, Morohashi T, Goto T. Evaluation of cold snare polypectomy for small pedunculated (Ip) polyps with thin stalks: a prospective clinical feasibility study. Scand J Gastroenterol. 2022 Feb;57(2):253-259. doi: 10.1080/00365521.2021.1998603. Epub 2021 Nov 2. PMID 34727817
- [Background] Arimoto J, Chiba H, Ashikari K, Fukui R, Tachikawa J, Okada N, Suto T, Kawano N, Niikura T, Kuwabara H, Nakaoka M, Ida T, Goto T, Nakajima A. Management of Less Than 10-mm-Sized Pedunculated (Ip) Polyps with Thin Stalk: Hot Snare Polypectomy Versus Cold Snare Polypectomy. Dig Dis Sci. 2021 Jul;66(7):2353-2361. doi: 10.1007/s10620-020-06436-7. Epub 2020 Jul 4. PMID 32623550
- [Background] Arimoto J, Chiba H, Ashikari K, Fukui R, Tachikawa J, Suto T, Kawano N, Niikura T, Kuwabara H, Nakaoka M, Ida T, Higurashi T, Goto T, Nakajima A. Safety and efficacy of cold snare polypectomy for pedunculated (Ip) polyps measuring less than 10 mm in diameter. Int J Colorectal Dis. 2020 May;35(5):859-867. doi: 10.1007/s00384-020-03547-5. Epub 2020 Feb 28. PMID 32112197
- [Background] Ferlitsch M, Hassan C, Bisschops R, Bhandari P, Dinis-Ribeiro M, Risio M, Paspatis GA, Moss A, Libanio D, Lorenzo-Zuniga V, Voiosu AM, Rutter MD, Pellise M, Moons LMG, Probst A, Awadie H, Amato A, Takeuchi Y, Repici A, Rahmi G, Koecklin HU, Albeniz E, Rockenbauer LM, Waldmann E, Messmann H, Triantafyllou K, Jover R, Gralnek IM, Dekker E, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2024. Endoscopy. 2024 Jul;56(7):516-545. doi: 10.1055/a-2304-3219. Epub 2024 Apr 26. PMID 38670139
- [Background] Tseng CH, Chang LC, Wu JL, Chang CY, Chen CY, Chen PJ, Shun CT, Hsu WF, Chen YN, Chen CC, Huang TY, Tu CH, Chen MJ, Chou CK, Lee CT, Chen PY, Lin JT, Wu MS, Chiu HM. Bleeding Risk of Cold Versus Hot Snare Polypectomy for Pedunculated Colorectal Polyps Measuring 10 mm or Less: Subgroup Analysis of a Large Randomized Controlled Trial. Am J Gastroenterol. 2024 Nov 1;119(11):2233-2240. doi: 10.14309/ajg.0000000000002847. Epub 2024 May 9. PMID 38775310